CLINICAL TRIAL: NCT01029522
Title: A Multi-center, Randomized, Double-blinded Equivalence Clinical Trial to Evaluate Efficacy and Safety of LipiLou 20 mg Versus Lipitor 20 mg in Hypercholesterolemic Patients With Higher Risk Cardiovascular Disease in Korea
Brief Title: Dyslipidemia in Cardiovascular Disease
Acronym: KoLipilou
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 224CHL08F
Record Dates: First submitted 2009-11-16; First posted 2009-12-10 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Dyslipidemia
Keywords: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lipilou 20mg (Experimental)
  Interventions: Drug: Atorvastatin (Lipilou)
- Lipitor 20mg (Active Comparator)
  Interventions: Drug: Atorvastatin (Lipitor)

INTERVENTIONS:
Drug: Atorvastatin (Lipilou) — treatment of dyslipidemia administration : PO, qod
  Arms: Lipilou 20mg
Drug: Atorvastatin (Lipitor) — treatment of dyslipidemia administration : PO, qod
  Other Names: Lipitor
  Arms: Lipitor 20mg

SUMMARY:
A multi-center, randomized, double-blinded equivalence clinical trial to evaluate efficacy and safety of LipiLou 20 mg versus Lipitor 20 mg in hypercholesterolemic patients with higher risk cardiovascular disease in Korea.

ELIGIBILITY:
Inclusion Criteria:

1. Dyslipidemic patients with high-risk cardiovascular disease meeting more than 1 requirement below (LDL-C ≥ 100mg/dL) 1) Coronary artery disease

   * diagnosed with atheroma in Coronary CT or Angiography, or SPECT positive or Treadmill test positive 2) Diabetes Mellitus 3) intervened with stent in coronary artery disease more than 1 year before 4) diagnosed with atheroma in carotid artery 5) Peripheral artery disease
2. Aged 20~85 years
3. Volunteers consented with participating clinical trial and submitted consent paper

Exclusion Criteria:

1. Experimental examination at screening 1) Active liver disease or more than 2 x ULN of AST/ALT 2) Creatine Kinase > 2 x ULN 3) Creatinine > 2.5mg/dL 4) Triglycerides > 500mg/dL
2. intervened with stent in coronary artery disease less than 1 year before
3. Hyper-sensitive or resistant to other HMG-CoA reductase inhibitors, or experienced serious adverse events
4. Patients taking dyslipidemic treatments within 4 weeks (HMG-CoA reductase inhibitors, fibrates, nicotinic acids or bile acid resins, etc.)
5. As uncontrolled DM patients, HbA1c≥11% or fasting plasma glucose ≥200mg/dL
6. DBP > 100mmHg, SBP > 160mmHg
7. Diagnosed with myopathy
8. Appear to be a risk of myopathy below

   * renal impairment or prior renal dysfunction
   * hypothyroidism
   * genetic defects or family history of myopathy
   * experienced prior muscle toxicity with taking statins or fibrates
   * prior liver disease or higher intakes of alcohol
   * aged over 70, and a risk of myopathy
9. Women pregnant or breast-feeding
10. Women capable of pregnancy without using contraceptives
11. contra-indicated medically or mentally, or forbidden legally
12. Enrolled to other clinical trial within 4 weeks
13. Impossible to participate clinical trial according to investigator's decision

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2008-08; Primary Completion 2008-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
LDL-C | after taken medicine for 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: KIM hyo soo, ph D, Principal Investigator — yongon-dong, jong-ro gu, Seoul National University Hospital, South of Korea